CLINICAL TRIAL: NCT07255716
Title: Postoperative Infections and Immune Profiles in Patients Undergoing LVAD Implantation
Status: Active, not recruiting | Type: Observational
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Collaborators: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2023CXGC011
Record Dates: First submitted 2025-11-20; First posted 2025-12-01 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Infection; Driveline Heart-assisted Device Related Infection; Pneumonia; Sepsis
Keywords: lvad; infection
MeSH Terms: conditions — Infections; Pneumonia; Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Peripheral blood samples retained for flow cytometry and single-cell RNA sequencing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- group1: All patients who met the inclusion criteria for LVAD implantation
  Interventions: Other: none intervention

INTERVENTIONS:
Other: none intervention — none intervention

SUMMARY:
The objective of this study is to investigate the incidence of infection and changes in the immune profile following left ventricular assist device implantation. The primary aim is to elucidate the relationship between postoperative infection and immune alterations and to identify risk factors predictive of postoperative infection.

DETAILED DESCRIPTION:
1. Background: left ventricular assist devices (LVADs) implantation is an important treatment for end-stage heart failure. Previous studies have indicated that implantation of a left ventricular assist device may alter a patient's immune status by affecting immune cells, which may be a significant reason for the high postoperative infection rate among patients. Previous studies have indicated that left ventricular assist device implantation may alter patients' immune status by affecting immune cells, which may be a significant factor contributing to high postoperative infection rates. The aim of this study is to evaluate infection events following LVAD implantation and their relationship with patients' immune status. this will be crucial for predicting infection occurrence and identifying potential intervention strategies.
2. Study design:

   Design Type: Retrospective, observational, multi-center study Study Population: patients who received LVAD implantations between June 2020 and October 2025 at 2 centers in China.

   Primary Objective: To evaluate the incidence of infection rate after LVAD implantation .

   Secondary Objectives: To identify factors associated with infection, assess the immune status alteration after LVAD implantation.
3. Study Population Inclusion criteria (i) age >18 years, (ii) indication for LVAD implantation, (iii)informed consent.

Exclusive criteria included active preoperative infection and no other circulatory support devices were used preoperatively

4. Data Collection

1. Demographic and clinical characteristics from medical records, including age, sex, comorbidities, heart failure etiologies, INTERMACS profiles.
2. Surgical details, including device type, duration of support, and concomitant surgeries.
3. Infection prevention measures, including the use of prophylactic antibiotics, skin decolonization procedures, driveline fixation sutures, etc.
4. Clinical examination data, including blood tests, imaging studies, cardiac function tests, etc.
5. Regular follow-up data, including clinical blood tests, changes in cardiac function, and incidence of infection events, along with collection of peripheral blood for assessment of immune status.

5. Statistical Analysis Descriptive statistics will be used to summarize patient demographics, infection incidence, and outcomes. Subgroup analyses will be conducted based on the types of postoperative infections.

Longitudinal clinical examination data were analyzed using longitudinal linear mixed models, with appropriate post-hoc comparisons via the emmeans package, applying Bonferroni adjustment for multiple testing.

Statistical significance will be indicated by the specific p-values for each comparison.

6. Expected Outcomes and Significance Primary Outcome: Incidence of different types of infections after LVAD implantation.

Secondary Outcomes: the longitudinal changes in immune indicators after LVAD implantation and the association between infection incidence and immune status.

The findings of this study may offer guidance for the clinical management of postoperative infections and support the development of potential intervention strategies.

7. Timeline Study Period: June 2020 to October 2025 Data Analysis Period: November 2024 to January 2025

ELIGIBILITY:
Inclusion Criteria:

(i) age >18 years, (ii) indication for LVAD implantation, (iii)informed consent.

Exclusion Criteria:

(i) active preoperative infection (ii) other circulatory support devices were used preoperatively

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving LVAD implantation who meet the inclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2025-11-15 (Actual); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
culture-proven infections | Infection confirmed within 90 days postoperatively is defined as early infection; infection confirmed after 90 days postoperatively is defined as late infection.

SECONDARY OUTCOMES:
immune parameters changes after LVAD implantation. | Blood test results available at various follow-up intervals from preoperative to postoperative periods, including 2 weeks, 1 month, 3 months, 6 months, etc.
  the longitudinal changes in clinical and immune parameters after LVAD implantation

CONTACTS AND LOCATIONS:
Locations (1):
- Fuwai Hospital, Beijing, Xicheng, China